CLINICAL TRIAL: NCT04178291
Title: Erythritol Powder Air Polishing as an Adjunct in Non-surgical Periodontal Therapy in the Management of Periodontitis: a Randomised Clinical Trial
Brief Title: Air Polishing as an Adjunct in Non-surgical Periodontal Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Nor Adinar Baharuddin, Associate Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101269-4
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Periodontitis
Keywords: Periodontitis; air polishing; randomised clinical trial; adjunct; debridement
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional debridement and air polishing (Experimental): All participants will receive full mouth EPAP as an adjunct to RSD using ultrasonic scalers and Gracey currettes. The EPAP procedure will be performed using the Air-Flow Master R (EMS) equipment. For supragingival biofilm removal, the Air-Flow handpiece will be used, while the Perio-Flow handpiece with a disposable nozzle will be used for subgingival debridement at sites with PPD ≥ 5mm. No time limit is applicable for supragingival air polishing. However, for subgingival debridement, the nozzle will be inserted for 5 seconds into each pocket, and moved vertically up and down. Gracey currettes will be used at sites with PPD ≥ 5mm.
  Interventions: Device: Ultrasonic scaler and Gracey currettes; Device: Air polishing with erythritol powder
- Conventional debridement (Active Comparator): All participants will receive full mouth RSD using ultrasonic scalers and Gracey currettes. Gracey currettes will be used at sites with PPD ≥ 5mm.
  Interventions: Device: Ultrasonic scaler and Gracey currettes

INTERVENTIONS:
Device: Ultrasonic scaler and Gracey currettes — Full mouth subgingival debridement using ultrasonic scaler and Gracey currettes
Device: Air polishing with erythritol powder — Air flow PLUS
  Arms: Conventional debridement and air polishing

SUMMARY:
Periodontal disease is an infection that causes inflammation and destruction of the tooth supporting structures, and if untreated, will eventually lead to tooth loss. Periodontal disease has been identified as a significant contributor to the global burden of oral disease. This disease is reported to be the sixth most prevalent disease globally. Periodontal disease has an association with diabetes, cardiovascular diseases and preterm low birth weight babies. Therefore, treatment of this disease is necessary. Treatment of periodontal disease involves mechanical removal of oral biofilm. Biofilm removal is initially carried out via non-surgical periodontal therapy, with subgingival debridement being one of the most important steps. According to the first European Workshop on Periodontology, subgingival debridement comprises subgingival instrumentation to disrupt and remove the oral biofilm. Subgingival debridement involves various techniques including hand instrumentation and ultrasonic instrumentation. Recently, treatment modality such as air polishing is also gaining momentum. Air polishing was reported to be more comfortable than conventional periodontal therapy. Besides, a number of studies had portrayed similar clinical outcomes with the use of air polishing in comparison to conventional periodontal therapy. However, there is no study evaluating the health economic aspect of these treatment modalities. Health economic evaluation is a valuable evaluation in intervention studies. Such evaluations provide information on the best way of using available resources in health care settings. For instance, advances in health care technology have resulted in an array of alternative treatment options. Unfortunately, such options tend to cost more than the existing therapeutic approaches. Therefore, economic evaluations will identify the worth of the new treatment options in comparison to the gold standard, in this case, comparing the adjunctive use of air polishing with conventional periodontal therapy. Besides focusing at patient reported outcomes and cost effectiveness of air polishing, this prospective, parallel, single-blinded, randomised controlled clinical trial is also planned to investigate the clinical and biological responses after the adjunct use of Erythritol Powder Air Polishing (EPAP) in addition to root surface debridement (RSD).

DETAILED DESCRIPTION:
Periodontal disease is an infection that causes inflammation of the tooth supporting structures, which results in the destruction of the periodontal ligament and alveolar bone, and eventually, tooth loss. The aetiology of the disease is oral biofilm. Therefore, the regular mechanical removal of biofilm, among others, is necessary to prevent and stop the disease progression. Biofilm and biofilm retentive calculus are removed via periodontal debridement. Subgingival debridement is an important procedure that is initially performed in the non-surgical periodontal therapy phase. According to the first European Workshop on Periodontology, subgingival debridement involves gently instrumenting subgingivally to disrupt and/or remove the biofilm. Various techniques are involved in subgingival debridement, with hand instruments and ultrasonic or sonic instruments being the most common, while modalities like air polishing are gaining momentum.

Mechanical periodontal debridement using hand instruments like curettes, sickles, hoes or files, and power driven instruments such as sonic or ultrasonic scalers, is generally known as root surface debridement (RSD). This modality is considered to be the gold standard of periodontal therapy. The usage of hand instruments has been advocated for their efficiency and the fact that it allows tactile sensation and operator control. However, various drawbacks from these instruments have been noted. Hand instruments and scalers are both technique sensitive, time consuming, and may cause irreversible hard tissue damage when used regularly. Besides, anatomical variations such as grooves, concavities and enamel pearls as well as deep pockets and furcation involvement, can influence debridement quality. Since periodontal therapy is performed regularly, being time efficient, acceptable to patient, and causing minimal tissue damage are important determinants. As such, treatment that causes minimal abrasion to root surface while being highly effective in biofilm removal would be a preferable choice.

One such treatment is air polishing. Air polishing was introduced in 1945 for the purpose of cavity preparation. Over time, its use expanded to periodontal debridement. Stain and biofilm are removed by the abrasive "slurry" which is formed by mixing together pressurised air, a jet of water and a stream of small particles. Sodium bicarbonate was the only abrasive powder available from the late 1970s until 2004. It is non-toxic and water soluble, with a mean size of up to 250μm. It has been shown to be safe and efficient to be

used on intact enamel surfaces. However, due to its abrasiveness, it could not be used on demineralised enamel surfaces. A study showed that regardless of parameters such as working time, powder and water setting, working distance, and angulation of the handpiece, substantial damage to the root occurs from sodium bicarbonate, concluding that it is contraindicated for use in exposed root surfaces. In order to overcome this problem, glycine based powders were then produced. In the in vitro study showed that glycine powder proved to have low abrasiveness towards cementum and dentine, while being efficient at plaque removal. The powder had a mean particle size of 45μm - 60μm, and was 80% less abrasive compared to sodium bicarbonate. More recently, erythritol powders have been used in air polishing. Erythritol is a sugar alcohol that is non-toxic, chemically neutral, and water soluble, and has been widely used as an artificial sweetener and food additive. Due to comparable physical properties to glycine and chemical characteristics allowing binding of antiseptic substances, it has been suggested for subgingival biofilm removal. Moreover, a recent study has shown erythritol to have an inhibitory effect on some periodontal bacteria, including P. gingivalis.

Advancements in air polishing devices have also occurred, mainly involving a disposable nozzle design to access the periodontal pocket directly, thus allowing the abrasive slurry to be delivered into moderate-to-deep periodontal pockets. The nozzle has a thickness of 0.7mm, which is within the diameter range of most periodontal probes, thereby allowing it to be inserted to the base of the pocket with minimal force. Besides, the new design resulted in a drop of pressure of the jet spray by 1 bar, thus reducing the risk of emphysema and allowing the nozzle to be used subgingivally.

The usage of air polishing in supportive periodontal therapy (SPT) has been extensively studied. However, minimal studies on the adjunctive use of air polishing in the management of active periodontitis have been conducted. One such study studied demonstrated that the effect of adjunctive subgingival glycerine powder air polishing (GPAP) in chronic periodontitis. It was a single blinded, 6 month study using the split mouth design with one of the outcomes being the reduction in the volume of gingival crevicular fluid (GCF). RSD followed by flushing of pockets with water was carried out in the control group, while RSD was followed by GPAP in the test group. Both groups showed significant reduction in periodontal parameters, and no significant differences between the two groups were seen. The test group showed significant reduction in GCF volume compared to control at 3 months, although at 6 months, no difference between the two groups was noted. Since GCF volume is an objective measure of subclinical inflammation, this study suggested that GPAP as an adjunct to RSD may improve periodontal inflammation in the short term.

Another study by Park et al. aimed to identify the clinical and microbiological effects of adjunctive subgingival erythritol powder air polishing (EPAP) in initial therapy. It was a 3 month study using a split mouth design in which treatment for the test group involved RSD and subgingival EPAP, whereas only RSD was done in the control group. Both groups showed significant changes in clinical parameters, and no difference was seen between the groups. Total bacterial count between baseline and 1 month after treatment decreased in both groups, but the decrease was significant in the test group. Between 1 month and 3 months after treatment, total bacterial count increased in both groups, but the increase was more significant in the control group. It appears that supplementing RSD with EPAP may have an effect on the total bacterial count. EPAP was also noted to have an anti-microbial effect, since the P. gingivalis count after 1 month treatment was significantly lower in the test group. This study concluded that both modes of treatment were clinically and microbiologically effective for initial therapy.

However, both studies were conducted using a split mouth design. Such a design has a risk of crossover effects, thus limiting intra-individual comparisons as local therapy can have systemic effects that are able to influence outcomes in different sites in the same individual. Therefore, there is a need to conduct a study using the parallel mouth design to identify the effects of adjunctive use of air polishing in periodontitis patient. Nevertheless, with new and more expensive technology, the question of cost effectiveness is not uncommon. Resources in health care such as time, money, and materials are often limited. This necessitates health economic evaluations to be carried out. One such evaluation is a cost effectiveness analysis that identifies the relationship between incremental resource consumption and outcome gain for various interventions. No such study has been conducted with regards to the cost effectiveness of air polishing. Therefore, the aim of this study is to investigate the adjunctive use of EPAP in NSPT and determine its cost effectiveness in the management of periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30-65 years old
2. Healthy or well controlled systemic diseases, including diabetes (HbA1c<7%) and hypertension (BP<140/90 mm Hg)
3. Diagnosed with moderate to severe periodontitis (Stage II and III) regardless of grade (Caton et al. 2017)
4. >20 remaining teeth

Exclusion Criteria:

1. Systemic conditions requiring antibiotic prophylaxis
2. Pregnant or breast feeding women
3. Immunosuppressive therapy
4. Immunocompromised such as HIV/AIDS patients
5. Periodontal therapy in the last 6 months
6. Antibiotic or anti-inflammatory therapy in the last 4 months
7. Known hypersensitivity to sugar alcohol (polyol)
8. Physical limitations or restrictions that prevent normal oral hygiene procedures
9. Heavy smoker who smokes ≥ 1 pack of cigarettes per day
10. Plaque score > 30%
11. Probing pocket depth > 6mm

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Changes in probing pocket depth (PPD). | 6 months
  Probing Pocket Depth (PPD) at 6 sites: Distance of margin of free gingiva to base of the pocket measured in millimetre using UNC-15 periodontal probe.

SECONDARY OUTCOMES:
Changes in clinical attachment level | 6 month
  To determine change in clinical attachment level, measured in millimetre, from cementoenamel junction to base of pocket (sum of periodontal pocket and recession).
Changes in recession | 6 month
  Gingival recession (REC): Distance from CEJ to margin of free gingiva measured in millimetre using UNC-15 periodontal probe.
Changes in Periodontal inflamed surface area | 6 months
  To determine change in periodontal inflamed surface area i.e. the sum of the periodontal pocket depth of bleeding on probing - positive sites for the total dentition and can be easily calculated using routine periodontal charting
Changes in full mouth bleeding score | 6 months
  Full mouth bleeding score (FMBS): Using Gingival Bleeding Index (Ainamo and Bay, 1975), bleeding will be assessed at 6 sites each tooth using a dichotomous scoring method. It will be considered as present (1) if there is bleeding within 10 seconds after probing of the gingiva, and absent (0) if there is no bleeding.
Changes in full mouth plaque score | 6 months
  Full mouth plaque score (FMPS): Using the Visible Plaque Index (Ainamo and Bay, 1975) visible plaque on the mesiobuccal, midbuccal, distobuccal, and lingual/palatal, surfaces will be recorded using a dichotomous scoring method. It will be considered as present (1) if there is visible plaque on the respective surfaces, and absent (0) if there is no visible plaque. Plaque disclosing solution will be used to aid in the scoring.
The ratio value of incremental Cost Effectiveness | 6 months
  Using Incremental Cost Effectiveness ratio to identify if the adjunctive use of air polishing during conventional periodontal treatment in periodontal pockets up to 6mm deep is cost effective compared to conventional periodontal therapy alone. The analytic horizon will be for six months.

CONTACTS AND LOCATIONS:
Locations (1):
- Nor Adinar Baharuddin, Kuala Lumpur, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savage A, Eaton KA, Moles DR, Needleman I. A systematic review of definitions of periodontitis and methods that have been used to identify this disease. J Clin Periodontol. 2009 Jun;36(6):458-67. doi: 10.1111/j.1600-051X.2009.01408.x. PMID 19508246
- [Background] Moene R, Decaillet F, Andersen E, Mombelli A. Subgingival plaque removal using a new air-polishing device. J Periodontol. 2010 Jan;81(1):79-88. doi: 10.1902/jop.2009.090394. PMID 20059420
- [Background] Laleman I, Cortellini S, De Winter S, Rodriguez Herrero E, Dekeyser C, Quirynen M, Teughels W. Subgingival debridement: end point, methods and how often? Periodontol 2000. 2017 Oct;75(1):189-204. doi: 10.1111/prd.12204. PMID 28758304
- [Background] Ng E, Byun R, Spahr A, Divnic-Resnik T. The efficacy of air polishing devices in supportive periodontal therapy: A systematic review and meta-analysis. Quintessence Int. 2018;49(6):453-467. doi: 10.3290/j.qi.a40341. PMID 29700503
- [Background] Lindhe J, Westfelt E, Nyman S, Socransky SS, Haffajee AD. Long-term effect of surgical/non-surgical treatment of periodontal disease. J Clin Periodontol. 1984 Aug;11(7):448-58. doi: 10.1111/j.1600-051x.1984.tb01344.x. PMID 6378986
- [Background] Kocher T, Fanghanel J, Sawaf H, Litz R. Substance loss caused by scaling with different sonic scaler inserts--an in vitro study. J Clin Periodontol. 2001 Jan;28(1):9-15. doi: 10.1034/j.1600-051x.2001.280102.x. PMID 11142673
- [Background] Flemmig TF, Petersilka GJ, Mehl A, Hickel R, Klaiber B. The effect of working parameters on root substance removal using a piezoelectric ultrasonic scaler in vitro. J Clin Periodontol. 1998 Feb;25(2):158-63. doi: 10.1111/j.1600-051x.1998.tb02422.x. PMID 9495615
- [Background] Ritz L, Hefti AF, Rateitschak KH. An in vitro investigation on the loss of root substance in scaling with various instruments. J Clin Periodontol. 1991 Oct;18(9):643-7. doi: 10.1111/j.1600-051x.1991.tb00104.x. PMID 1960232
- [Background] Zappa U, Smith B, Simona C, Graf H, Case D, Kim W. Root substance removal by scaling and root planing. J Periodontol. 1991 Dec;62(12):750-4. doi: 10.1902/jop.1991.62.12.750. PMID 1765938
- [Background] Leknes KN. The influence of anatomic and iatrogenic root surface characteristics on bacterial colonization and periodontal destruction: a review. J Periodontol. 1997 Jun;68(6):507-16. doi: 10.1902/jop.1997.68.6.507. PMID 9203093
- [Background] Petersilka GJ. Subgingival air-polishing in the treatment of periodontal biofilm infections. Periodontol 2000. 2011 Feb;55(1):124-42. doi: 10.1111/j.1600-0757.2010.00342.x. No abstract available. PMID 21134232
- [Background] Kontturi-Narhi V, Markkanen S, Markkanen H. Effects of airpolishing on dental plaque removal and hard tissues as evaluated by scanning electron microscopy. J Periodontol. 1990 Jun;61(6):334-8. doi: 10.1902/jop.1990.61.6.334. PMID 2366141
- [Background] Petersilka GJ, Bell M, Mehl A, Hickel R, Flemmig TF. Root defects following air polishing. J Clin Periodontol. 2003 Feb;30(2):165-70. doi: 10.1034/j.1600-051x.2003.300204.x. PMID 12622860
- [Background] Petersilka GJ, Bell M, Haberlein I, Mehl A, Hickel R, Flemmig TF. In vitro evaluation of novel low abrasive air polishing powders. J Clin Periodontol. 2003 Jan;30(1):9-13. doi: 10.1034/j.1600-051x.2003.300102.x. PMID 12702105
- [Background] Munro IC, Berndt WO, Borzelleca JF, Flamm G, Lynch BS, Kennepohl E, Bar EA, Modderman J. Erythritol: an interpretive summary of biochemical, metabolic, toxicological and clinical data. Food Chem Toxicol. 1998 Dec;36(12):1139-74. doi: 10.1016/s0278-6915(98)00091-x. PMID 9862657
- [Background] Hagi TT, Hofmanner P, Salvi GE, Ramseier CA, Sculean A. Clinical outcomes following subgingival application of a novel erythritol powder by means of air polishing in supportive periodontal therapy: a randomized, controlled clinical study. Quintessence Int. 2013 Nov-Dec;44(10):753-61. doi: 10.3290/j.qi.a30606. PMID 24078975
- [Background] Hashino E, Kuboniwa M, Alghamdi SA, Yamaguchi M, Yamamoto R, Cho H, Amano A. Erythritol alters microstructure and metabolomic profiles of biofilm composed of Streptococcus gordonii and Porphyromonas gingivalis. Mol Oral Microbiol. 2013 Dec;28(6):435-51. doi: 10.1111/omi.12037. Epub 2013 Jul 29. PMID 23890177
- [Background] Flemmig TF, Arushanov D, Daubert D, Rothen M, Mueller G, Leroux BG. Randomized controlled trial assessing efficacy and safety of glycine powder air polishing in moderate-to-deep periodontal pockets. J Periodontol. 2012 Apr;83(4):444-52. doi: 10.1902/jop.2011.110367. Epub 2011 Aug 23. PMID 21861637
- [Background] Garnick JJ, Silverstein L. Periodontal probing: probe tip diameter. J Periodontol. 2000 Jan;71(1):96-103. doi: 10.1902/jop.2000.71.1.96. PMID 10695944
- [Background] Tsang YC, Corbet EF, Jin LJ. Subgingival glycine powder air-polishing as an additional approach to nonsurgical periodontal therapy in subjects with untreated chronic periodontitis. J Periodontal Res. 2018 Jun;53(3):440-445. doi: 10.1111/jre.12532. Epub 2018 Mar 25. PMID 29574763
- [Background] Park EJ, Kwon EY, Kim HJ, Lee JY, Choi J, Joo JY. Clinical and microbiological effects of the supplementary use of an erythritol powder air-polishing device in non-surgical periodontal therapy: a randomized clinical trial. J Periodontal Implant Sci. 2018 Oct 24;48(5):295-304. doi: 10.5051/jpis.2018.48.5.295. eCollection 2018 Oct. PMID 30405937
- [Background] Antczak-Bouckoms AA, Tulloch JF, Berkey CS. Split-mouth and cross-over designs in dental research. J Clin Periodontol. 1990 Aug;17(7 Pt 1):446-53. doi: 10.1111/j.1600-051x.1990.tb02343.x. PMID 2201705
- [Background] Listl S, Birch S. Reconsidering value for money in periodontal treatment. J Clin Periodontol. 2013 Apr;40(4):345-8. doi: 10.1111/jcpe.12085. No abstract available. PMID 23488994
- [Background] Mohd-Dom TN, Wan-Puteh SE, Muhd-Nur A, Ayob R, Abdul-Manaf MR, Abdul-Muttalib K, Aljunid SM. Cost-Effectiveness of Periodontitis Management in Public Sector Specialist Periodontal Clinics: A Societal Perspective Research in Malaysia. Value Health Reg Issues. 2014 May;3:117-123. doi: 10.1016/j.vhri.2014.04.012. Epub 2014 May 20. PMID 29702916
- [Background] Christodoulides N, Nikolidakis D, Chondros P, Becker J, Schwarz F, Rossler R, Sculean A. Photodynamic therapy as an adjunct to non-surgical periodontal treatment: a randomized, controlled clinical trial. J Periodontol. 2008 Sep;79(9):1638-44. doi: 10.1902/jop.2008.070652. PMID 18771363
- See also: Glossary — https://www.ncbi.nlm.nih.gov/mesh/?term=periodontal+debridement